CLINICAL TRIAL: NCT00521183
Title: Translational Phase I Trial of Escalating Doses of 5-Chloro-2'-Deoxycytidine (CldC) With a Fixed Dose of Tetrahydrouridine Combined With External Brain Radiation for Metastatic Carcinoma to the Brain
Brief Title: Cytochlor, Tetrahydrouridine, and External-Beam Radiation Therapy in Treating Patients With Cancer That Has Spread to the Brain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Brian Lally (Other)
Responsible Party: Sponsor-Investigator, Brian Lally, Assistant Professor of Clinical, University of Miami
Organization: University of Miami (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20057104; SCCC-2005097 (Other: University of Miami Sylvester Comprehensive Cancer Center); WIRB-20051340 (Other: Western Institutional Review Board)
Record Dates: First submitted 2007-08-24; First posted 2007-08-27 (Estimated); Last update posted 2014-11-25 (Estimated); Status verified 2014-11

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult tumors metastatic to brain
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms | interventions — Centers for Disease Control and Prevention, U.S.; Tetrahydrouridine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CldC + H4U (Experimental)
  Interventions: Drug: Cytochlor; Drug: Tetrahydrouridine; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Cytochlor — The study's starting dose of CldC is 50 mg/m2/day. The dose of CldC will be escalated / de-escalated for patients. Patients will receive CldC+H4U on 3 days (Wed, Thr, Fri) in week 1, which precedes the initiation of radiation therapy. Patients will receive H4U and CldC IV by bolus infusion. Treatment with CldC+H4U will then continue for 5 days (Mon-Fri) during each of weeks 2 and 3, and will be accompanied by radiation therapy at 3 Gy/fraction initiated 3-4 h after bolus infusion of CldC+H4U. Treatment with CldC+H4U and radiation will then stop at the end of week 3.
  Other Names: CldC, CDC
Drug: Tetrahydrouridine — A fixed dose of H4U at 720 mg/m2/day will be used, regardless of the dose of CldC administered. H4U will be delivered by an IV bolus infusion over a period of 5 minutes, followed 5 minutes later by an IV bolus infusion of CldC. Patients will receive CldC+H4U on 3 days (Wed, Thr, Fri) in week 1, which precedes the initiation of radiation therapy. Patients will receive H4U and CldC IV by bolus infusion. Treatment with CldC+H4U will then continue for 5 days (Mon-Fri) during each of weeks 2 and 3, and will be accompanied by radiation therapy at 3 Gy/fraction initiated 3-4 h after bolus infusion of CldC+H4U. Treatment with CldC+H4U and radiation will then stop at the end of week 3.
  Other Names: THU, H4U
Radiation: Radiation Therapy — One treatment of 3 Gy will be given daily 5 days per week (10 fractions) for a total of 30 Gy over two weeks.

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Drugs, such as cytochlor and tetrahydrouridine, may make tumor cells more sensitive to radiation therapy.

PURPOSE: This phase I trial is studying the side effects and best dose of cytochlor when given together with tetrahydrouridine and external-beam radiation therapy in treating patients with cancer that has spread to the brain.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Establish the safety and toxicity profile of cytochlor and H4U when given in combination with external-beam radiotherapy for 2 weeks after treatment with the drugs alone in the previous week.

Secondary

* Determine the effectiveness of H4U to inhibit systemic cytidine deaminase (CD) during the course of treatment with cytochlor and H4U.
* Perform detailed pharmacokinetic studies to determine the levels of cytochlor and its metabolites in serum and in urine in weeks 1, 2, and 3 during treatment.

OUTLINE: This is a dose-escalation study of cytochlor.

Patients receive cytochlor IV and tetrahydrouridine (H4U) IV over 5 minutes on 3 days in week 1 and on days 1-5 in weeks 2 and 3. Patients also undergo external-beam radiotherapy 5 days a week in weeks 2 and 3 initiated 3-4 hours after infusions of cytochlor and H4U. Treatment may repeat in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed monthly for 3 months, every 3 months for 1 year, every 4 months for 1 year, every 6 months for 1 year, and then yearly thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of metastatic cancer to the brain by contrast-enhanced MRI or CT scan
* Eligible for whole-brain radiotherapy (WBRT)

  * Patients treated with prior surgery are eligible if WBRT is to be used post operatively
  * Not planning to be treated with stereotactic radiosurgery
* No leptomeningeal metastasis documented by contrast-enhanced MRI/CT scan or cerebrospinal fluid evaluation

PATIENT CHARACTERISTICS:

Inclusion criteria:

* Karnofsky performance status (PS) 70-100% or ECOG PS 0-1
* Leukocytes ≥ 3,000/µL
* Absolute neutrophil count > 1,500/µL
* Platelet count > 100,000/µL
* Total bilirubin normal
* AST and ALT < 2.5 times upper limit of normal
* Creatinine normal OR creatinine clearance > 60 mL/min
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation

Exclusion criteria:

* Uncontrolled intercurrent illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or lactating
* Alcohol dependence

PRIOR CONCURRENT THERAPY:

* No prior radiotherapy to the brain
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent chemotherapy, immunotherapy, hormonal therapy (excluding contraceptives and replacement steroids), or other experimental medication
* No other concurrent anticancer therapy outside the protocol

  * Systemic therapy one month before or after brain radiotherapy is allowed
* No concurrent heparin or coumadin

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2007-06; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
To establish a dose range of CldC for further clinical studies (Phase II clinical trials) based on safety and toxicity. | 2 Years
b) Establish the safety and toxicity profile of CldC+ H4U when given in combination with RT for 2 weeks following treatment with the drug alone for 3 days in the week prior to the combined treatment. | Duration of study treatment

SECONDARY OUTCOMES:
a) Determine the effectiveness of H4U to inhibit systemic cytidine deaminase (CD) during the course of treatment with CldC + H4U. | At protocol specified timepoints during treatment
  Baseline Levels of CD will be obtained by assaying CD in serum prior to initiation of treatment on Wednesday of week 1. Follow-up assays of CD in serum will be made on the Fridays of weeks 1 to 3 after each day's treatment with CldC + H4U. In weeks 2 and 3 this will take place prior to RT
Cytochlor and metabolite levels in serum at weeks 1, 2, and 3 | Pharmacokinetic sampling at protocol-specified timepoints during duration of treatment
Cytochlor and metabolite levels in urine at weeks 1, 2, and 3 | Pharmacokinetic sampling at protocol-specified timepoints during duration of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Fazilat Ishkanian, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States